CLINICAL TRIAL: NCT05522283
Title: Performance of Stool and Serum Cytomegalovirus Real-time Polymerase Chain Reaction and Their Combination in Diagnosing CMV Colitis
Brief Title: Stool and Serum CMV-PCR in Diagnosing CMV Colitis
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Julajak Limsrivilai, Principal Investigator, Mahidol University
Other Study IDs: Si 810/2020
Record Dates: First submitted 2022-08-27; First posted 2022-08-31 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: CMV Colitis
Keywords: Cytomegalovirus, CMV, PCR, Fecal, stool, serum, colitis
MeSH Terms: conditions — Cytomegalovirus Infections; Pathologic Complete Response; Colitis | interventions — Defecation; Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CMV colitis: Patients with the detection of either cytomegalic cells or IHC-CMV cells were diagnosed with CMV colitis.
  Interventions: Diagnostic Test: Stool and blood CMV PCR
- Non-CMV colitis: Symptomatic patients were not detected with either cytomegalic cells or IHC-CMV cells.
  Interventions: Diagnostic Test: Stool and blood CMV PCR
- Healthy volunteers: Asymptomatic patients underwent colonoscopy for screening.
  Interventions: Diagnostic Test: Stool and blood CMV PCR

INTERVENTIONS:
Diagnostic Test: Stool and blood CMV PCR — Quantitative stool CMV-PCR (CMV R-gene® kit, limit of detection 450 copies/ml, Biomerieux, France) and quantitative serum CMV-PCR (Cobas® CMV, limit of detection 150 copies/ml, Roche, USA) were collected within seven days of colonoscopy.
  Other Names: Colonoscopy with colonic tissue biopsy

SUMMARY:
CMV viral load detected by real-time polymerase chain reaction (PCR) in either serum or stool may be beneficial in diagnosing CMV colitis, but the data is limited. Therefore, we aimed to investigate the diagnostic performance of stool CMV-PCR, serum CMV-PCR, and their combination in diagnosing CMV colitis using tissue histopathology as the standard reference in patients with clinical suspicion of CMV colitis.

DETAILED DESCRIPTION:
The gold standard for diagnosing CMV colitis is colonoscopy with tissue biopsy. Histology by hematoxylin and eosin stain (H&E) has a high specificity of 92-100% but low sensitivity of 10-87%. Immunohistochemistry stain(IHC) increases diagnostic sensitivity to 78-93%.Tissue polymerase chain reaction assay (PCR), the method that amplifies CMV DNA, has the highest sensitivity (92-93%); however, there is no clear cut-off value to differentiate CMV bystanders from CMV colitis. Although colonoscopy is the gold standard, it is not permitted to be performed in some situations due to a high risk of procedural complications, such as in patients with profound neutropenia, thrombocytopenia, or severe illnesses. Serum CMV-PCR is a non-invasive test that detects CMV viremia, which could be associated with CMV-GI disease. However, the results of previous studies are inconsistent.

In recent years, there has been an increasing interest in stool CMV-PCR in diagnosing CMV colitis. Stool CMV-PCR is a non-invasive test that can be either qualitative or quantitative. In the first pilot study, Herfarth et al. reported stool CMV-PCR sensitivity of 83% and specificity of 93% in 19 inflammatory bowel disease patients. Since that, there have been only a few studies reporting the performance of stool CMV-PCR in diagnosing CMV colitis, and their results are inconsistent. The reported sensitivity ranges from 16.7% to 85%, and the specificity ranges from 71 to 96%. Furthermore, the diagnostic performance of combining serum and stool CMV-PCR, which could improve diagnostic performance, has not been studied. Therefore, we aimed to investigate the diagnostic performance of stool CMV-PCR, serum CMV-PCR, and their combination in diagnosing CMV colitis using tissue histopathology as the standard reference in patients with clinical suspicion of CMV colitis. In addition, we also evaluated the correlation of viral load in stool, serum, colonic tissue, and numbers of CMV-infected cells in colonic tissue.

Patients older than 18 years with clinical suspicion of CMV colitis were enrolled. The criteria for clinically suspicious of CMV colitis included: i) presence of at least one of the risk factors, including human immunodeficiency virus infection, solid organ or hematologic stem cell transplantations, hematologic malignancy, inflammatory bowel disease, taking immunosuppressive agents or chemotherapy, and critically ill with multiple comorbidities, and ii) presenting with gastrointestinal tract symptoms, including abdominal pain, gastrointestinal bleeding, diarrhea, and bowel ileus.

All participants underwent colonoscopy with tissue biopsy for both H&E stain and immunohistochemistry for CMV (IHC-CMV). Patients with the detection of either cytomegalic cells or IHC-CMV cells were diagnosed with CMV colitis. The other two pieces of colonic tissue were sent for quantitative CMV-PCR (CMV R-gene® kit, limit of detection 450 copies/ml, Biomerieux, France). Patients who could not proceed with the colonoscopy and tissue biopsy were excluded. Quantitative stool CMV-PCR (CMV R-gene® kit, limit of detection 450 copies/ml, Biomerieux, France) and quantitative serum CMV-PCR (Cobas® CMV, limit of detection 150 copies/ml, Roche, USA) were collected within seven days of colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with clinical suspicion of CMV colitis were enrolled.

Exclusion Criteria:

* Patients who could not proceed with the colonoscopy and tissue biopsy were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The criteria for clinically suspicious of CMV colitis included:
  i) presence of at least one of the risk factors, including human immunodeficiency virus infection, solid organ or hematologic stem cell transplantations, hematologic malignancy, inflammatory bowel disease, taking immunosuppressive agents or chemotherapy, and critically ill with multiple comorbidities, and ii) presenting with gastrointestinal tract symptoms, including abdominal pain, gastrointestinal bleeding, diarrhea, and bowel ileus
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of stool and serum CMV PCR | within 7 days of colonoscopy
  Sensitivity, specificity, and AOC in the diagnosis of CMV colitis

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology division, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sattayalertyanyong O, Limsrivilai J, Phaophu P, Subdee N, Horthongkham N, Pongpaibul A, Angkathunyakul N, Chayakulkeeree M, Pausawasdi N, Charatcharoenwitthaya P. Performance of Cytomegalovirus Real-Time Polymerase Chain Reaction Assays of Fecal and Plasma Specimens for Diagnosing Cytomegalovirus Colitis. Clin Transl Gastroenterol. 2023 May 1;14(5):e00574. doi: 10.14309/ctg.0000000000000574. PMID 36854054